CLINICAL TRIAL: NCT06770114
Title: A Clinical Study to Investigate a New Mouthwash Containing 0.075% CPC, and 0.1% Hyaluronic Acid and 0.28% Zinc Lactate as Compared to a Fluoride Mouthwash Containing 0.044% NaF in Reducing Plaque and Helping Prevent Gum Problems on Dental Implants Over a 6-month Period of Product Use
Brief Title: Clinical Study to Investigate a New Mouthwash in Reducing Plaque and Helping Prevent Gum Problems on Dental Implants Over a 6-month Period of Product Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRO-2021-12-PIM-IMW-ITA-YPZ
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Cetylpyridinium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- New Mouthwash containing CPC, Zinc and Hyaluronic acid (Experimental): After brushing in the morning and in the evening, 20 ml of mouthwash shall be used for each rinsing, 2 times daily (morning and evening ) for 30 seconds each time. No further rinsing with water shall be occurred after spilt out and after each mouthwash rising. Each qualified subject will follow this specific application for 6 months
  Interventions: Drug: Cetylpyridinium Chloride, Zinc Lactate and Hyaluronic Acid Mouthwash
- Fluoride Mouthwash (Active Comparator): After brushing in the morning, 10 ml of mouthwash shall be used for each rinsing, 1 time daily (morning ) for 60 seconds each time. No further rinsing with water shall be occurred after spilt out and after each mouthwash rising. Each qualified subject will follow this specific application for 6 months.
  Interventions: Drug: PhosFlur Mouthwash

INTERVENTIONS:
Drug: Cetylpyridinium Chloride, Zinc Lactate and Hyaluronic Acid Mouthwash — 0 .075 % cetylpyridinium chloride and 0 .28 % zinc lactate
  Arms: New Mouthwash containing CPC, Zinc and Hyaluronic acid
Drug: PhosFlur Mouthwash — 0 .044 % sodium fluoride
  Arms: Fluoride Mouthwash

SUMMARY:
The objective of this six-month clinical research study is to evaluate the clinical efficacy of a new mouthwash on helping prevent gum problems (gingival index scores ) in adults as compared to a control mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the six-month duration of the clinical research study.
* Good general health.
* Minimum of two dental implants (2 different quadrants ), each implant must have a restoration.
* Initial mucositis index of at least 1 .0 as determined by the use of the Mombelli Modified Gingival Index.
* Initial plaque index of at least 1 .5 as determined by the use of the Mombelli Modified Plaque Index.
* Signed Informed Consent Form.

Exclusion Criteria:

* Presence of orthodontic bands.
* Tumor (s ) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and /or extensive loss of periodontal attachment or alveolar bone ) or peri-implantitis.
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care /personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Self-reported pregnant or lactating subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Mombelli Modified Gingival Index | baseline
  Initial mucositis index of at least 1.0 as determined by the use of the Mombelli Modified Gingival
Mombelli Modified Gingival Index | three month
  Initial mucositis index of at least 1.0 as determined by the use of the Mombelli Modified Gingival
Mombelli Modified Gingival Index | six month
  Initial mucositis index of at least 1.0 as determined by the use of the Mombelli Modified Gingival
Mombelli Modified Plaque Index | baseline
  Initial plaque index of at least 1 .5 as determined by the use of the Mombelli Modified Plaque
Mombelli Modified Plaque Index | three month
  Initial plaque index of at least 1 .5 as determined by the use of the Mombelli Modified Plaque
Mombelli Modified Plaque Index | six month
  Initial plaque index of at least 1 .5 as determined by the use of the Mombelli Modified Plaque

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Montesani, DDS, Principal Investigator — University of Rome
Locations (1):
- Clinica Odontoiatrica Montesani, Roma, Rome, Italy